CLINICAL TRIAL: NCT00438204
Title: A Phase II Trial of Pemetrexed, Gemcitabine, and Bevacizumab Every Two Weeks in Chemotherapy-Naive Patients With Stages IIIB/IV Non- Squamous, Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Pemetrexed Disodium, Gemcitabine, and Bevacizumab in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: All data collection has completed.
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Antoinette J. Wozniak, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000531832; P30CA022453 (NIH); WSU-2005-008 (Other: Barbara Ann Karmanos Cancer Institute); WSU-036806MP4F (Other: Wayne State University - Human Investigation Committee)
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer; large cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Bevacizumab; Gemcitabine; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab, gemcitabine hydrochloride (Experimental): Bevacizumab 10mg/kg IV over 90 ± 15 minutes every 14 days
  Gemcitabine 1200 mg/m2 intravenously over 30 minutes following the pemetrexed disodium every 14 days
  Pemetrexed 400 mg/m2 intravenously over 10 minutes every 14 days.
  Interventions: Biological: bevacizumab; Drug: gemcitabine hydrochloride; Drug: pemetrexed disodium

INTERVENTIONS:
Biological: bevacizumab — Bevacizumab 10mg/kg IV over 90 ± 15 minutes every 14 days
  Other Names: Avastin ®
Drug: gemcitabine hydrochloride — Gemcitabine 1200 mg/m2 intravenously over 30 minutes following the pemetrexed every 14 days
  Other Names: Gemzar ®
Drug: pemetrexed disodium — Pemetrexed disodium 400 mg/m2 intravenously over 10 minutes every 14 days.
  Other Names: Alimta®

SUMMARY:
RATIONALE: Pemetrexed disodium may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving pemetrexed disodium and gemcitabine together with bevacizumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving pemetrexed disodium and gemcitabine together with bevacizumab works in treating patients with stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of pemetrexed disodium, gemcitabine hydrochloride, and bevacizumab in chemotherapy-naïve patients with stage IIIB or IV nonsquamous cell non-small cell lung cancer.

Secondary

* Determine the response rate in patients treated with this regimen.
* Determine the time to treatment failure in patients treated with this regimen.
* Determine the overall survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: Patients receive pemetrexed disodium IV over 10 minutes, gemcitabine hydrochloride IV over 30 minutes, and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 14 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients may then receive bevacizumab alone in the absence of disease progression or unacceptable toxicity.

After the completion of study treatment, patients are followed periodically for 6 months.

PROJECTED ACCRUAL: A total of 42 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria

* Histologic or cytologic proof of non-squamous non-small cell lung cancer (NSCLC) (adenocarcinoma, bronchioloalveolar, large cell carcinoma).
* Must have Stage IV or IIIB NSCLC. Patients with Stage IIIB must have a pleural effusion or not be candidates for treatment for locally advanced disease with chemoradiotherapy.
* Cannot have a tumor with cavitation..
* Have uni-dimensional measurable or evaluable disease. If disease is within a previous radiation port there must be documented progression.
* 18 years of age and have a life expectancy of greater than 12 weeks.
* Must not have had prior chemotherapy for advanced disease.
* Must have an ECOG performance status of 0-1.
* With treated brain metastases are eligble. for details.
* Adequate organ function:

Absolute neutrophil count of > 1.5 x 109/L Platelet count > 100,000/109/L Hemoglobin > 8g/dl Calculated creatinine clearance > 45mL/min using the standard Cockroft and Gault formula Hepatic: bilirubin < 1.5 times the upper limit of normal,alkaline phosphatase, aspartate transaminase (AST) and alanine transaminase (ALT) < 3 times upper limit of normal. Alkaline phosphatase, AST, ALT < 5 times upper limit of normal is acceptable if liver has tumor involvement. Urine protein:creatinine ratio ≤1.0 at screening

* Patients of reproductive potential must use an approved contraceptive method during and for 3 months after study.
* Must sign an informed consent that details the investigational nature of the study according to the institutional and federal guidelines.
* Registered with the clinical trials office of the institution.

Exclusion Criteria

* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study
* Prior chemotherapy except for erlotinib for advanced disease.
* Uncontrolled hypertension (Blood pressure of >150/100 mmHg )
* Unstable angina
* New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix E)
* History of myocardial infarction within 6 months prior to day 1
* History of hemorrhagic or thrombotic stroke or other CNS bleed within 6 months prior to day 1
* Clinically significant peripheral vascular disease of 61
* Evidence of bleeding diathesis or coagulopathy. Patients must not require full dose anticoagulants for any reason.
* Known CNS disease, except for treated brain metastasis Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to Day 0
* Urine protein:creatinine ratio > or = 1.0 at screening
* History of abdominal fistula, gastrointestinal perforation, or intraabdominal abscess within 6 months prior to Day 0
* Serious, non-healing wound, ulcer, or bone fracture
* Evidence of cavitation in the tumor.
* Intrathoracic lung carcinoma of squamous cell histology Mixed tumors will be categorized by the predominant cell type unless small cell elements are present, in which case the patient is ineligible; sputum cytology alone is unacceptable.
* Extrathoracic-only squamous cell NSCLC are eligible. Patients with only peripheral lung lesions (of any NSCLC histology) will also be eligible.
* History of hemoptysis (bright red blood of 1/2 teaspoon or more within 28 days of registration or clinical history of > Grade 2
* Clinically significant effusions that cannot be drained
* Inability to comply with study and/or follow-up procedures
* Previous or concurrent malignancies with the exception of adequately treated squamous cell or basal cell carcinoma of the skin, in situ carcinoma of the cervix, or any other malignancy treated and in clinical remission for more than 3 years.
* Prior radiation therapy to the target lesion, unless the lesion is clearly progressing and the interval between the most recent radiation therapy and enrollment is at least 4 weeks.
* Pregnancy or lactating females. All pre-menopausal women should have a negative urine pregnancy test prior to enrollment. All patients of reproductive potential should agree to use an effective contraceptive method.
* Serious concomitant systemic disorders (including oncologic emergencies) incompatible with the study (at the discretion of the investigator).
* Inability to interrupt non-steroidal anti-inflammatory agents 2 days before, the day of, and 2 days after the dose of pemetrexed.
* Disease which cannot be radiologically imaged.
* Inability to take dexamethasone, folic acid or vitamin B12 administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-05; Primary Completion 2013-03 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette J. Wozniak, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (2):
- United States (2):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab, Gemcitabine Hydrochloride: Bevacizumab 10mg/kg IV over 90 ± 15 minutes every 14 days
  Gemcitabine 1200 mg/m2 intravenously over 30 minutes following the pemetrexed every 14 days
  Pemetrexed 400 mg/m2 intravenously over 10 minutes every 14 days.
  bevacizumab: Bevacizumab 10mg/kg IV over 90 ± 15 minutes every 14 days
  gemcitabine hydrochloride: Gemcitabine 1200 mg/m2 intravenously over 30 minutes following the pemetrexed every 14 days
  pemetrexed disodium: Pemetrexed 400 mg/m2 intravenously over 10 minutes every 14 days.
Period: Overall Study
Arm/Group | Bevacizumab, Gemcitabine Hydrochloride
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab, Gemcitabine Hydrochloride
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: RECIST criteria for tumor progression of at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: Up to 12 months
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Bevacizumab, Gemcitabine Hydrochloride
Number analyzed (Participants) | 39
months | 6.1 [3.9 to 7.6]

2. Secondary Outcome: Number of Participants With Response
Description: The rate of response per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Every 8 weeks, for up to 54 months
Measure: Count of Participants; unit: Participants
Groups:
- Bevacizumab, Gemcitabine Hydrochloride: Bevacizumab 10mg/kg IV over 90 ± 15 minutes every 14 days
  Gemcitabine 1200 mg/m2 intravenously over 30 minutes following the pemetrexed disodium every 14 days
  Pemetrexed 400 mg/m2 intravenously over 10 minutes every 14 days.
  bevacizumab: Bevacizumab 10mg/kg IV over 90 ± 15 minutes every 14 days
  gemcitabine hydrochloride: Gemcitabine 1200 mg/m2 intravenously over 30 minutes following the pemetrexed every 14 days
  pemetrexed disodium: Pemetrexed disodium 400 mg/m2 intravenously over 10 minutes every 14 days.
Arm/Group | Bevacizumab, Gemcitabine Hydrochloride
Number analyzed (Participants) | 39
Participants
  Complete response | 1
  Partial response | 15
  Stable disease | 12
  Progressive disease | 10
  Not response evaluable | 1

3. Secondary Outcome: Number of Participants With Grade 3 or Grade 4 Toxicity
Description: Grade 3/4 toxicity according to the NCI Common Toxicity Criteria v3.0 .
Time Frame: Every two weeks, for up to 54 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab, Gemcitabine Hydrochloride
Number analyzed (Participants) | 39
Participants
  Neutropenia | 11
  Leukopenia | 3
  Anemia | 1
  Thrombocytopenia | 1
  Febrile Neutropenia | 1
  Elevated ALT/AST | 4
  Acute renal insufficiency | 1
  Anorexia | 2
  Thrombosis/embolism | 3
  Dehydration | 1
  Fatigue | 7
  Hyperglycemia | 9
  Hypertension | 2
  Nausea/vomiting | 1
  Bowel Perforation | 1
  Dyspnea | 4
  Diverticulitis | 2
  Ataxia | 1

4. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure using the Kaplan-Meier method.
Time Frame: Every 8 weeks, for up to 54 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab, Gemcitabine Hydrochloride
Number analyzed (Participants) | 39
months | 6.2 [3.9 to 8.0]

5. Secondary Outcome: Overall Survival
Description: Overall survival using the Kaplan-Meier method.
Time Frame: Every 8 weeks, for up to 54 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab, Gemcitabine Hydrochloride
Number analyzed (Participants) | 39
months | 17.5 [8.4 to 28.0]

ADVERSE EVENTS:
Time Frame: Approximately 7 years
Arm/Group | Bevacizumab, Gemcitabine Hydrochloride
Serious Adverse Events (participants affected / at risk) | 18/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab, Gemcitabine Hydrochloride (N=39)
Neutrophils (Investigations) | 11 (11)
White blood cells (WBC) (Investigations) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 4 (4)
Acute renal insufficiency (Renal and urinary disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Fatigue (General disorders) | 7 (7)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (9)
Hypertension (Vascular disorders) | 2 (2)
Hypophospatemia (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness-generalized (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Bowel Perforation (Gastrointestinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Right otitis media (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Perforation (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 3 (3)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Neutropenia (Metabolism and nutrition disorders) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Pancytopenia (Investigations) | 1 (1)
Pulmonary Embolism (Vascular disorders) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Right side pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab, Gemcitabine Hydrochloride (N=39)
WBC (Investigations) | 21 (21)
Hgb (Blood and lymphatic system disorders) | 32 (32)
ANC (Investigations) | 12 (12)
Platelets (Investigations) | 3 (3)
Fatigue (General disorders) | 24 (24)
Fever (General disorders) | 9 (9)
Rash (Skin and subcutaneous tissue disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 13 (13)
Diarrhea (Gastrointestinal disorders) | 9 (9)
Vomiting (Gastrointestinal disorders) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 12 (12)
Aspartate aminotransferase (AST) increased (Investigations) | 13 (13)
Alanine Aminotransferase (ALT) increased (Investigations) | 14 (14)
Hyperglycemia (Metabolism and nutrition disorders) | 24 (24)
Hypertension (Vascular disorders) | 11 (11)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Muscle weakness-generalized (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 10 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Alkaline Phosphotase increased (Investigations) | 5 (5)
Creatinine increased (Investigations) | 4 (4)
Proteinuria (Renal and urinary disorders) | 10 (10)
Fluid retention syndrome (FRS) (Musculoskeletal and connective tissue disorders) | 9 (9)
Pain (General disorders) | 14 (14)
Infrection systemic (Infections and infestations) | 6 (6)
Lung hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
There were no significant limitations of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No